CLINICAL TRIAL: NCT00112437
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, and Efficacy of MK-0822 (Cathepsin K Inhibitor) in the Treatment of Postmenopausal Women With Osteoporosis
Brief Title: A Study to Examine the Effects of an Experimental Drug on Postmenopausal Osteoporosis (MK-0822-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-004; 2005_023
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2010-05-13 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2017-12

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — odanacatib; Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium Carbonate; Drug: Placebo
- Odanacatib 3 mg (Experimental)
  Interventions: Drug: Odanacatib; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium Carbonate
- Odanacatib 10 mg (Experimental)
  Interventions: Drug: Odanacatib; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium Carbonate
- Odanacatib 25 mg (Experimental)
  Interventions: Drug: Odanacatib; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium Carbonate
- Odanacatib 50 mg (Experimental)
  Interventions: Drug: Odanacatib; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium Carbonate

INTERVENTIONS:
Drug: Odanacatib — Odanacatib 3 mg, once weekly for 24 months
  Other Names: MK-0822
  Arms: Odanacatib 3 mg
Drug: Odanacatib — Odanacatib 10 mg, once weekly for 24 months
  Other Names: MK-0822
  Arms: Odanacatib 10 mg
Drug: Odanacatib — Odanacatib 25 mg, once weekly for 24 months
  Other Names: MK-0822
  Arms: Odanacatib 25 mg
Drug: Odanacatib — Odanacatib 50 mg, once weekly for 24 months
  Other Names: MK-0822
  Arms: Odanacatib 50 mg
Dietary Supplement: Vitamin D3 — Vitamin D3, two 2800 IU weekly throughout the study
Dietary Supplement: Calcium Carbonate — Participants who have a calcium intake less than 1000 mg/day will receive daily calcium supplements providing 500 mg of elemental calcium.
Drug: Placebo — Placebo to Odanacatib 3 mg, 10 mg, 25 mg, or 50 once weekly for 24 months
  Arms: Placebo

SUMMARY:
This is a 1-year base study with a 1-year extension to examine the effects of a new experimental medication (odanacatib [MK-0822]) on postmenopausal osteoporosis. This study will enroll approximately 375 postmenopausal women, and randomly assign them to 4 different doses of odanacatib or to placebo. Measurements performed during the study include: bone mineral density scans, spine x-rays, laboratory blood and urine tests, height measurements and optional bone biopsies (at the end of 2 years).

DETAILED DESCRIPTION:
Study Extension:

Participants who completed 12 months of the base study and 12 months of the first extension were invited to continue in three additional extensions: MK0-822-004-10, which extended the study to 36 months, MK-0822-004-20 (NCT00112437) which extended the study to 60 months, and MK-0822-004-30 (NCT00112437), which extended the study to 120 months.

* In the first extension, participants continued to receive the same treatment they received in the 12-month base study.
* In the second extension, participants were re-randomized to odanacatib 50 mg OW or placebo OW for 12 months.
* In the third extension, participants who were initially randomized to odanacatib 3 mg or placebo OW in the base study received odanacatib 50 mg weekly in Years 4 and 5; all other participants remained on the same treatment they were during Year 3.
* In the fourth extension, all participants received odanacatib weekly in Years 6-10.

Study arms for extensions include only odanacatib 50 mg and placebo for the first two extensions and odanacatib 50 mg only for the third extension.

Extension Studies:

MK-0822-004-10 (NCT00112437) Extension: Participant has participated in and completed 24 months of treatment in the base study

MK-0822-004-20 (NCT00112437) Extension: Participant participated in and completed 36 months of treatment in base and extension studies.

MK-0822-004-30 (NCT00112437) Extension: Participant participated in and completed 60 months of treatment in the base and extension studies.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal for 5 or more years, defined as no menses for at least 5 years OR at least 5 years status post bilateral oophorectomy
* Bone mineral density T-score at the hip or spine of -2.0 or less
* Spinal anatomy suitable for dual-energy x-ray absorptiometry (DXA). At the lumbar spine, there is no evidence of vertebral fracture in at least 3 vertebrae in the L1 to L4 region on baseline spine films. (Significant scoliosis, bony trauma, degenerative joint disease, and sequelae of orthopedic procedures that result in anatomy that is unsuitable for accurate bone densitometry must be absent from the lumbar spine.)
* At least one hip must be evaluable by DXA (e.g., contain no hardware from orthopedic procedures)
* In a state of general health allowing for successful completion of the trial
* Agreement to not use any medications to treat osteoporosis during the study

Exclusion Criteria:

* History of prior osteoporotic fracture (unless declined treatment with or was ineligible for osteoporosis therapy)
* Past treatment with osteoporosis medications, steroids, hormone replacement, as well as various other medications that affect bone may be exclusionary. (Different exclusion criteria apply to each bone active drug. For example, any prior use of intravenous (IV) bisphosphonates is not permitted. By contrast, prior use of hormone replacement for several years is permitted if it has not occurred within the past 6 months. Please ask the study doctor for details)
* Significant clinical or laboratory abnormalities at the screening visit for the study that, in the opinion of the investigator, could complicate interpretation of the study results or pose additional risk to the patient (for example, patients who are non-ambulatory should be excluded for this reason)

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2005-06-24 (Actual); Primary Completion 2007-12-26 (Actual); Study Completion 2016-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Bone HG, McClung MR, Roux C, Recker RR, Eisman JA, Verbruggen N, Hustad CM, DaSilva C, Santora AC, Ince BA. Odanacatib, a cathepsin-K inhibitor for osteoporosis: a two-year study in postmenopausal women with low bone density. J Bone Miner Res. 2010 May;25(5):937-47. doi: 10.1359/jbmr.091035. PMID 19874198
- [Result] Langdahl B, Binkley N, Bone H, Gilchrist N, Resch H, Rodriguez Portales J, Denker A, Lombardi A, Le Bailly De Tilleghem C, Dasilva C, Rosenberg E, Leung A. Odanacatib in the treatment of postmenopausal women with low bone mineral density: five years of continued therapy in a phase 2 study. J Bone Miner Res. 2012 Nov;27(11):2251-8. doi: 10.1002/jbmr.1695. PMID 22777865
- [Result] Rizzoli R, Benhamou CL, Halse J, Miller PD, Reid IR, Rodriguez Portales JA, DaSilva C, Kroon R, Verbruggen N, Leung AT, Gurner D. Continuous treatment with odanacatib for up to 8 years in postmenopausal women with low bone mineral density: a phase 2 study. Osteoporos Int. 2016 Jun;27(6):2099-107. doi: 10.1007/s00198-016-3503-0. Epub 2016 Feb 15. PMID 26879200
- [Derived] Eisman JA, Bone HG, Hosking DJ, McClung MR, Reid IR, Rizzoli R, Resch H, Verbruggen N, Hustad CM, DaSilva C, Petrovic R, Santora AC, Ince BA, Lombardi A. Odanacatib in the treatment of postmenopausal women with low bone mineral density: three-year continued therapy and resolution of effect. J Bone Miner Res. 2011 Feb;26(2):242-51. doi: 10.1002/jbmr.212. PMID 20740685

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 375 participants were recruited from June 2005 to December 2005. Investigators used one or more of the following recruitment methods: Investigator Patient/Subject Database or Medical Records, Investigator's Local Recruitment/Advertising, Other Health Professional and, Physician Referral (Primary/Specialist/Family Doctor).
Pre-assignment Details: Participants entered screening followed by a 3-week placebo run-in. All took vitamin D3, 5600 IU once weekly, those with average daily calcium intakes <1000 mg took calcium 500 mg/day as calcium carbonate. Participants were excluded from the active treatment based on predetermined exclusion criteria (Bone Mineral Density and laboratory results).
Groups:
- Placebo-Base; Placebo-Ext 1: One placebo tablet once a week
- Odanacatib 3 Mg-Base; Odanacatib 3 Mg-Ext 1: One odanacatib 3 mg tablet once a week
- Odanacatib 10 Mg-Base; Odanacatib 10 Mg-Ext 1: One odanacatib 10 mg tablet once a week
- Odanacatib 25 Mg-Base; Odanacatib 25 Mg-Ext 1: One odanacatib 25 mg tablet once a week
- Odanacatib 50 Mg-Base; Odanacatib 50 Mg-Ext 1: One odanacatib 50 mg tablet once a week
- Placebo / Placebo-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one placebo tablet once a week. Before entering this extension, participants in this treatment group had taken one placebo tablet once a week for 2 years.
- Placebo / Odanacatib 50 Mg-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one 50 mg tablet of odanacatib once a week. Before entering this extension, participants in this treatment group had taken one placebo tablet once a week for 2 years.
- Odanacatib 3 mg / Placebo-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one placebo tablet once a week. Before entering this extension, participants in this treatment group had taken one 3 mg tablet of odanacatib once a week for 2 years.
- Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one 50 mg tablet of odanacatib once a week. Before entering this extension, participants in this treatment group had taken one 3 mg tablet of odanacatib once a week for 2 years.
- Odanacatib 10 mg / Placebo-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one placebo tablet once a week. Before entering this extension, participants had taken one 10 mg tablet of odanacatib once a week for 2 years.
- Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one 50 mg tablet of odanacatib once a week. Before entering this extension, participants in this treatment group took one 10 mg tablet of odanacatib once a week for 2 years.
- Odanacatib 25 mg / Placebo-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one placebo tablet once a week. Before entering this extension, participants in this treatment group had taken one 25 mg tablet of odanacatib once a week for 2 years.
- Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one 50 mg tablet of odanacatib once a week. Before entering this extension, participants in this treatment group had taken one 25 mg tablet of odanacatib once a week for 2 years.
- Odanacatib 50 mg / Placebo-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one placebo tablet once a week. Before entering this extension, participants in this treatment group had taken one 50 mg tablet of odanacatib once a week for 2 years.
- Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one 50 mg tablet of odanacatib once a week. Before entering this extension, participants in this treatment group had taken one 50 mg tablet of odanacatib once a week for 2 years.
- Placebo Once Weekly-Ext 3: During this 24-month extension (Years 4-5), participants in this treatment group received one placebo tablet once a week.
- Odanacatib 50 mg Once Weekly-Ext 3: During this 24-month extension (Years 4-5), participants in this treatment group received one odanacatib 50 mg tablet once a week.
- Group A: Odanacatib 50 mg Once Weekly-Ext 4: During this 60-month extension (Years 6-10), participants in this treatment group received one odanacatib 50 mg tablet one a week. Group A consisted of a combination of participants who were treated with odanacatib 25 mg for 2 years,then odanacatib 50 mg for 8 years; and participants who were treated with odanacatib 50 mg for 10 years.
- Group B: Odanacatib 50 mg Once Weekly-Ext 4: During this 60-month extension (Years 6-10), participants in this treatment group received one odanacatib 50 mg tablet one a week. Group B consisted of a combination participants who were treated with placebo for 2 years, then odanacatib 50 mg for 8 years; participants who were treated with odanacatib 3 mg for 2 years, then odanacatib 50 mg for 8 years; and participants who were treated with odanacatib 10 mg for 2 years, then odanacatib 50 mg for 8 years.
- Group C: Odanacatib 50 mg Once Weekly-Ext 4: During this 60-month extension (Years 6-10), participants in this treatment group received one odanacatib 50 mg tablet one a week. Group C consisted of a combination of participants who were treated with placebo for 3 years, then odanacatib 50 mg for 7 years; and participants who were treated with odanacatib 3 mg for 2 years, then placebo for 1 year, then odanacatib 50 mg for 7 years.
- Group D: Odanacatib 50 mg Once Weekly-Ext 4: During this 60-month extension (Years 6-10), participants in this treatment group received one odanacatib 50 mg tablet once a week. Group D consists of a combination of participants who were treated with odanacatib 10 mg for 2 years, then placebo for 3 years, then odanacatib 50 mg for 5 years; participants who were treated with odanacatib 25 mg for 5 years, then placebo for 3 years, then odanacatib 50 mg for 5 years; and participants who were treated with odanacatib 50 mg for 2 years, then placebo for 3 years, then odanacatib 50 mg for 5 years.
Period: Year 1 (12-Month Base Study)
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1 | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / Placebo-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2 | Placebo Once Weekly-Ext 3 | Odanacatib 50 mg Once Weekly-Ext 3 | Group A: Odanacatib 50 mg Once Weekly-Ext 4 | Group B: Odanacatib 50 mg Once Weekly-Ext 4 | Group C: Odanacatib 50 mg Once Weekly-Ext 4 | Group D: Odanacatib 50 mg Once Weekly-Ext 4
Started | 83 | 82 | 77 | 79 | 78 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 68 (1 patient completed base study after December 19, 2006 and is not included in completed total.) | 64 (1 patient completed base study after December 19, 2006 and is not included in completed total.) | 65 | 71 | 66 (1 patient completed base study after December 19, 2006 and is not included in the completed total.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 15 | 18 | 12 | 8 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 9 | 10 | 6 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 5 | 2 | 1 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — moved | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — patient was unsure that they needed drug | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — DXA was lower by more than 8% | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Year 2 (12-Month Extension)
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1 | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / Placebo-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2 | Placebo Once Weekly-Ext 3 | Odanacatib 50 mg Once Weekly-Ext 3 | Group A: Odanacatib 50 mg Once Weekly-Ext 4 | Group B: Odanacatib 50 mg Once Weekly-Ext 4 | Group C: Odanacatib 50 mg Once Weekly-Ext 4 | Group D: Odanacatib 50 mg Once Weekly-Ext 4
Started | 0 | 0 | 0 | 0 | 0 | 63 | 62 | 63 | 69 | 63 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 60 | 53 | 55 | 62 | 50 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 9 | 8 | 7 | 13 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 6 | 1 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Patient stopped taking medication | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — patient was out of windows | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Moved | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Year 3 (12-Month Extension)
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1 | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / Placebo-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2 | Placebo Once Weekly-Ext 3 | Odanacatib 50 mg Once Weekly-Ext 3 | Group A: Odanacatib 50 mg Once Weekly-Ext 4 | Group B: Odanacatib 50 mg Once Weekly-Ext 4 | Group C: Odanacatib 50 mg Once Weekly-Ext 4 | Group D: Odanacatib 50 mg Once Weekly-Ext 4
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 22 | 18 | 17 | 18 | 17 | 19 | 21 | 18 | 20 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 17 | 18 | 16 | 17 | 13 | 16 | 20 | 16 | 19 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 0 | 1 | 1 | 4 | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — cortisone therapy, upcoming surgery | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Years 4-5 (24-Month Extension)
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1 | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / Placebo-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2 | Placebo Once Weekly-Ext 3 | Odanacatib 50 mg Once Weekly-Ext 3 | Group A: Odanacatib 50 mg Once Weekly-Ext 4 | Group B: Odanacatib 50 mg Once Weekly-Ext 4 | Group C: Odanacatib 50 mg Once Weekly-Ext 4 | Group D: Odanacatib 50 mg Once Weekly-Ext 4
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 100 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 37 | 92 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 8 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Discontinued for other reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Participant moved | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Period: Years 6-10 (60-Month Extension)
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1 | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / Placebo-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2 | Placebo Once Weekly-Ext 3 | Odanacatib 50 mg Once Weekly-Ext 3 | Group A: Odanacatib 50 mg Once Weekly-Ext 4 | Group B: Odanacatib 50 mg Once Weekly-Ext 4 | Group C: Odanacatib 50 mg Once Weekly-Ext 4 | Group D: Odanacatib 50 mg Once Weekly-Ext 4
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28 | 34 | 23 | 32
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 22 | 22 | 27
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 12 | 1 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base | Total
Number analyzed (Participants) | 83 | 82 | 77 | 79 | 78 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (7.8) | 63.1 (7.3) | 64.5 (8.0) | 62.9 (7.4) | 64.5 (8.1) | 64.2 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 82 | 77 | 79 | 78 | 399
  Male | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at 12 Months
Description: Percentage change in lumbar spine BMD (relative to baseline) at 12 Months.
Time Frame: Baseline and 12 months
Population: Analysis at Month 12 used Full-Analysis-Set Population of participants who took at least one dose of study medication and had necessary follow-up information, in their randomization treatment group, with last observation data carried forward. Seven patients had a baseline value, but no value at Month 12 for lumbar spine Bone Mineral Density.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base
Number analyzed (Participants) | 81 | 79 | 77 | 78 | 77
Percentage change | -0.13 [-0.80 to 0.54] | -0.62 [-1.30 to 0.05] | 1.50 [0.82 to 2.19] | 2.65 [1.97 to 3.33] | 3.37 [2.68 to 4.05]
Statistical Analysis 1: Comparison: Placebo-Base vs Odanacatib 50 Mg-Base; The primary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on lumbar spine BMD compared to placebo over 12 months. The primary hypothesis states that odanacatib will increase lumbar spine BMD compared to placebo over 12 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — Significance for the primary endpoint was achieved through stepdown trend-test, the highest dose group was removed and the test was repeated until lack of significance was observed; Stepwise linear trend test on ANCOVA model with treatment (scales 0, 1, 2, 3, 4) as covariate and center as factor in the model, with 5% significance; Difference in Least Squares Means = 3.50, 95% CI 2-sided [2.54 to 4.45]
Statistical Analysis 2: Comparison: Placebo-Base vs Odanacatib 25 Mg-Base; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 2.78, 95% CI 2-sided [1.82 to 3.73]
Statistical Analysis 3: Comparison: Placebo-Base vs Odanacatib 10 Mg-Base; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 1.63, 95% CI 2-sided [0.68 to 2.59]
Statistical Analysis 4: Comparison: Placebo-Base vs Odanacatib 3 Mg-Base; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.343, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.49, 95% CI 2-sided [-1.44 to 0.46]

2. Primary Outcome: Percentage Change From Baseline in Lumbar Spine BMD at 24 Months
Description: Percentage change in lumbar spine BMD (relative to baseline) at 24 Months.
Time Frame: Baseline and 24 months
Population: Analysis on lumbar spine BMD (g/cm2) at Month 24 used the Full-Analysis-Set Population with Last Observation Carried Forward from Month 18 to 24. No data were carried forward from the core to the extension period. Only patients who took at least one dose of extension medication were included. 17 patients were excluded from FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1
Number analyzed (Participants) | 62 | 58 | 60 | 65 | 58
Percentage Change | -0.19 [-1.13 to 0.75] | -1.03 [-2.00 to -0.07] | 3.20 [2.25 to 4.15] | 4.26 [3.35 to 5.18] | 5.48 [4.52 to 6.44]
Statistical Analysis 1: Comparison: Placebo-Ext 1 vs Odanacatib 50 Mg-Ext 1; The primary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on lumbar spine BMD compared to placebo over 24 months. The primary hypothesis states that odanacatib will increase lumbar spine BMD compared to placebo over 24 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 5.67, 95% CI 2-sided [4.32 to 7.02]
Statistical Analysis 2: Comparison: Placebo-Ext 1 vs Odanacatib 25 Mg-Ext 1; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 4.45, 95% CI 2-sided [3.15 to 5.76]
Statistical Analysis 3: Comparison: Placebo-Ext 1 vs Odanacatib 10 Mg-Ext 1; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 3.39, 95% CI 2-sided [2.06 to 4.73]
Statistical Analysis 4: Comparison: Placebo-Ext 1 vs Odanacatib 3 Mg-Ext 1; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.218, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Square Means = -0.84, 95% CI [-2.19 to 0.51]

3. Secondary Outcome: Percentage Change From Baseline in Total Hip BMD at 12 Months
Description: Percentage change in total hip BMD (relative to baseline) at 12 months
Time Frame: Baseline and 12 months
Population: This analysis was performed at Month 12 using Full-Analysis-Set approach with Last Observation Carried Forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base
Number analyzed (Participants) | 81 | 79 | 77 | 78 | 77
Percentage Change | -0.61 [-1.22 to -0.01] | -1.36 [-1.97 to -0.75] | 1.05 [0.44 to 1.67] | 1.45 [0.84 to 2.07] | 1.87 [1.25 to 2.49]
Statistical Analysis 1: Comparison: Placebo-Base vs Odanacatib 50 Mg-Base; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on total hip BMD compared to placebo over 12 months. The secondary hypothesis states that odanacatib will increase total hip BMD compared to placebo over 12 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — Significance for secondary endpoints was only declared if there was also significance for the primary endpoint. Multiplicity was addressed through a stepdown trend-test approach. Multiplicity for multiple endpoints was handled by a Hochberg procedure; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 2.49, 95% CI 2-sided [1.62 to 3.35]
Statistical Analysis 2: Comparison: Placebo-Base vs Odanacatib 25 Mg-Base; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 2.06, 95% CI 2-sided [1.20 to 2.93]
Statistical Analysis 3: Comparison: Placebo-Base vs Odanacatib 10 Mg-Base; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 1.67, 95% CI 2-sided [0.80 to 2.53]
Statistical Analysis 4: Comparison: Placebo-Base vs Odanacatib 3 Mg-Base; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.135, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.75, 95% CI 2-sided [-1.61 to 0.11]

4. Secondary Outcome: Percentage Change From Baseline in Femoral Neck BMD at 12 Months
Description: Percentage change in femoral neck BMD (relative to baseline) at 12 months
Time Frame: Baseline and 12 months
Population: This analysis was performed at Month 12 using Full-Analysis-Set approach with Last Observation Carried Forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base
Number analyzed (Participants) | 81 | 79 | 77 | 78 | 77
Percentage change | -0.13 [-0.79 to 0.54] | -0.32 [-0.99 to 0.35] | 0.74 [0.05 to 1.42] | 1.76 [1.08 to 2.44] | 2.53 [1.85 to 3.21]
Statistical Analysis 1: Comparison: Placebo-Base vs Odanacatib 50 Mg-Base; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on femoral neck BMD compared to placebo over 12 months. The secondary hypothesis states that odanacatib will increase femoral neck BMD compared to placebo over 12 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 2.66, 95% CI 2-sided [1.71 to 3.61]
Statistical Analysis 2: Comparison: Placebo-Base vs Odanacatib 25 Mg-Base; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — Significance for secondary endpoints was only declared if there was also significance for the primary endpoint. Multiplicity was addressed through stepdown trend-test approach. Multiplicity for multiple endpoints was handled by a Hochberg procedure; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 1.89, 95% CI 2-sided [0.93 to 2.84]
Statistical Analysis 3: Comparison: Placebo-Base vs Odanacatib 10 Mg-Base; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.095, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 0.87, 95% CI 2-sided [-0.09 to 1.82]
Statistical Analysis 4: Comparison: Placebo-Base vs Odanacatib 3 Mg-Base; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.19, 95% CI 2-sided [-1.14 to 0.75]

5. Secondary Outcome: Percentage Change From Baseline in Trochanter BMD at 12 Months
Description: Percentage change in trochanter BMD (relative to baseline) at 12 months
Time Frame: Baseline and 12 Months
Population: This analysis was performed at Month 12 using Full-Analysis-Set approach with Last Observation Carried Forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base
Number analyzed (Participants) | 81 | 79 | 77 | 78 | 77
Percentage change | -0.73 [-1.64 to 0.18] | -1.02 [-1.94 to -0.10] | 1.65 [0.72 to 2.58] | 1.91 [0.99 to 2.84] | 2.21 [1.28 to 3.14]
Statistical Analysis 1: Comparison: Placebo-Base vs Odanacatib 50 Mg-Base; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on trochanter BMD compared to placebo over 12 months. The secondary hypothesis states that odanacatib will increase trochanter BMD compared to placebo over 12 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 2.94, 95% CI 2-sided [1.64 to 4.24]
Statistical Analysis 2: Comparison: Placebo-Base vs Odanacatib 25 Mg-Base; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 2.65, 95% CI 2-sided [1.35 to 3.94]
Statistical Analysis 3: Comparison: Placebo-Base vs Odanacatib 10 Mg-Base; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 2.38, 95% CI 2-sided [1.08 to 3.69]
Statistical Analysis 4: Comparison: Placebo-Base vs Odanacatib 3 Mg-Base; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.731, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.29, 95% CI 2-sided [-1.58 to 1.00]

6. Secondary Outcome: Percentage Change From Baseline in Total Body BMD at 12 Months
Description: Percentage change in total body BMD (relative to baseline) at 12 months
Time Frame: Baseline and 12 Months
Population: This analysis was performed at Month 12 using Full-Analysis-Set Population with Last Observation Carried Forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base
Number analyzed (Participants) | 72 | 71 | 70 | 75 | 70
Percentage change | -0.42 [-1.16 to 0.32] | -1.89 [-2.64 to -1.14] | -1.06 [-1.81 to -0.30] | -0.51 [-1.23 to 0.22] | -0.13 [-0.89 to 0.62]
Statistical Analysis 1: Comparison: Placebo-Base vs Odanacatib 50 Mg-Base; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on total body BMD compared to placebo over 12 months. The secondary hypothesis states that odanacatib will increase total body BMD compared to placebo over 12 months; Test type: Superiority or Other; p = 0.112, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 0.29, 95% CI 2-sided [-0.77 to 1.35]
Statistical Analysis 2: Comparison: Placebo-Base vs Odanacatib 25 Mg-Base; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; ANCOVA — Significance for secondary endpoints was only declared if there was also significance for the primary endpoint. Multiplicity was addressed through a stepdown trend-test approach. Multiplicity for multiple endpoints was handle by a Hochberg procedure; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.09, 95% CI 2-sided [-1.13 to 0.95]
Statistical Analysis 3: Comparison: Placebo-Base vs Odanacatib 10 Mg-Base; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.63, 95% CI 2-sided [-1.69 to 0.42]
Statistical Analysis 4: Comparison: Placebo-Base vs Odanacatib 3 Mg-Base; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.47, 95% CI 2-sided [-2.53 to -0.42]

7. Secondary Outcome: Percentage Change From Baseline in Distal Forearm BMD at 12 Months
Description: Percentage change in distal forearm BMD (relative to baseline) at 12 months
Time Frame: Baseline and 12 Months
Population: This analysis was performed at Month 12 using Full-Analysis-Set Population with Last Observation Carried Forward
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base
Number analyzed (Participants) | 81 | 79 | 77 | 78 | 77
Percentage change | -1.27 [-1.98 to -0.57] | -2.55 [-3.26 to -1.83] | -1.00 [-1.73 to -0.28] | -0.17 [-0.89 to 0.55] | -0.04 [-0.77 to 0.68]
Statistical Analysis 1: Comparison: Placebo-Base vs Odanacatib 50 Mg-Base; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on distal forearm BMD compared to placebo over 12 months. The secondary hypothesis states that odanacatib will increase distal forearm BMD compared to placebo over 12 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 1.23, 95% CI 2-sided [0.22 to 2.24]
Statistical Analysis 2: Comparison: Placebo-Base vs Odanacatib 25 Mg-Base; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.005, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 1.10, 95% CI 2-sided [0.09 to 2.11]
Statistical Analysis 3: Comparison: Placebo-Base vs Odanacatib 10 Mg-Base; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.630, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 0.27, 95% CI 2-sided [-0.74 to 1.29]
Statistical Analysis 4: Comparison: Placebo-Base vs Odanacatib 3 Mg-Base; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -1.27, 95% CI 2-sided [-2.28 to -0.27]

8. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Urinary N-Telopeptides of Type I Collagen [u-NTx]) at 12 Months
Description: Back-transformation (geometric mean) of the Least Squares (LS) Mean of the log-values Percentage change from baseline, in Biochemical Marker of Bone turnover (urinary N-telopeptides of Type I collagen (u-NTx)) at 12 Months
Time Frame: Baseline and 12 Months
Population: This analysis was geometric mean percent change from baseline (which is a back-transformation of a log-transformed fraction from baseline) at Month 12 using a Per-Protocol approach. Participants with important protocol deviations and major protocol violators were excluded from the analyses. The per-protocol approach did not estimate missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base
Number analyzed (Participants) | 62 | 57 | 56 | 63 | 56
Percentage change | -2.37 [-14.78 to 11.85] | 8.80 [-5.50 to 25.27] | -34.21 [-42.94 to -24.15] | -48.29 [-54.80 to -40.84] | -60.23 [-65.51 to -54.13]
Statistical Analysis 1: Comparison: Placebo-Base vs Odanacatib 50 Mg-Base; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on biochemical indices of bone resorption (u-NTx) compared to placebo over 12 months. The secondary hypothesis states that odanacatib will decrease biochemical indices of bone resorption (u-NTx) over 12 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Stepwise linear trend test on ANCOVA model of log-fraction with treatment (scales 0, 1, 2, 3, 4) as covariate and center as factor, 5% significance; Difference in Least Squares Means = -57.86, 95% CI 2-sided [-72.33 to -43.38] — Difference in Least Squares Means (back-transformation of difference in log-fractions from baseline)
Statistical Analysis 2: Comparison: Placebo-Base vs Odanacatib 25 Mg-Base; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -45.92, 95% CI 2-sided [-60.93 to -30.91] — Difference in Least Squares Means (back-transformation of difference in log-fractions from baseline)
Statistical Analysis 3: Comparison: Placebo-Base vs Odanacatib 10 Mg-Base; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -31.84, 95% CI 2-sided [-48.11 to -15.58] — Difference in Least Squares Means (back-transformation of difference in log-fractions from baseline)
Statistical Analysis 4: Comparison: Placebo-Base vs Odanacatib 3 Mg-Base; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.249, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = 11.17, 95% CI 2-sided [-0.94 to 43.24] — Difference in Least Squares Means (back-transformation of difference in log-fractions from baseline)

9. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Serum C-Telopeptides of Type 1 Collagen [s-CTx]) at 12 Months
Description: Back-transformation (geometric mean) of the Least Squares (LS) Mean of the log-values Percentage change from baseline in Biochemical Marker of Bone turnover (serum C-telopeptides of Type 1 collagen (s-CTx)) at 12 Months.
Time Frame: Baseline and 12 Months
Population: This analysis was a geometric mean percent change from baseline (which is a back-transformation of a log-transformed fraction from baseline) at Month 12 using a Per-Protocol approach. Participants with important protocol deviations and major protocol violators were excluded from the analyses. The Per-Protocol approach did not estimate missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base
Number analyzed (Participants) | 62 | 57 | 56 | 62 | 55
Percentage change | -0.58 [-16.79 to 18.78] | 19.12 [-0.94 to 43.24] | -22.24 [-35.45 to -6.32] | -36.15 [-46.54 to -23.75] | -56.91 [-64.31 to -47.99]
Statistical Analysis 1: Comparison: Placebo-Base vs Odanacatib 50 Mg-Base; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on biochemical indices of bone resorption (s-CTx) compared to placebo over 12 months. The secondary hypothesis states that odanacatib will decrease biochemical indices of bone resorption (s-CTx) over 12 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -56.33, 95% CI [-75.86 to -36.81] — Difference in Least Squares Means (back-transformation from difference in log-fraction)
Statistical Analysis 2: Comparison: Placebo-Base vs Odanacatib 25 Mg-Base; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = -35.57, 95% CI [-56.63 to -14.51] — Difference in Least Square Means (back-transformation from difference in log-fraction)
Statistical Analysis 3: Comparison: Placebo-Base vs Odanacatib 10 Mg-Base; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.080, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -21.66, 95% CI [-44.54 to 1.23] — Difference in Least Squares Means (back-transformation from difference in log-fraction)
Statistical Analysis 4: Comparison: Placebo-Base vs Odanacatib 3 Mg-Base; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = 19.70, 95% CI 2-sided [-8.48 to 47.88] — Difference in Least Squares Means (back-transformation from difference in log-fraction)

10. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Urinary Total Deoxypyridinolines [u-DPyr]) at 12 Months
Description: Back-transformation (geometric mean) of the Least Squares Mean of the log-values percentage change from baseline in biochemical marker of bone turnover (urinary total deoxypyridinolines (u-DPyr)) (relative to baseline) at 12 Months
Time Frame: Baseline and 12 months
Population: This analysis was a geometric mean percent change from baseline (back-transformation of a log-transformed fraction from baseline) at Month 12 using a Per-Protocol approach. Participants with important protocol deviations and major protocol violators were excluded from the analyses. The per-protocol approach did not estimate missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base
Number analyzed (Participants) | 60 | 57 | 55 | 63 | 55
Percentage change | -7.25 [-19.73 to 7.18] | 20.91 [4.33 to 40.12] | -8.58 [-21.33 to 6.24] | -8.50 [-20.52 to 5.33] | -25.52 [-35.93 to -13.43]
Statistical Analysis 1: Comparison: Placebo-Base vs Odanacatib 50 Mg-Base; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on biochemical indices of bone resorption (u-DPyr) compared to placebo over 12 months. The secondary hypothesis states that odanacatib will decrease biochemical indices of bone resorption (u-DPyr) over 12 months; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -18.28, 95% CI 2-sided [-35.82 to -0.74] — Difference in Least Squares Means (back-transformation of difference in log-fractions from baseline)
Statistical Analysis 2: Comparison: Placebo-Base vs Odanacatib 25 Mg-Base; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.344, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -1.26, 95% CI 2-sided [-19.90 to 17.39] — Difference in Least Squares Means (back-transformation of difference in log-fractions from baseline)
Statistical Analysis 3: Comparison: Placebo-Base vs Odanacatib 10 Mg-Base; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -1.33, 95% CI 2-sided [-20.55 to 17.89] — Difference in Least Squares Means (back-transformation of difference in log-fractions from baseline)
Statistical Analysis 4: Comparison: Placebo-Base vs Odanacatib 3 Mg-Base; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = 28.15, 95% CI 2-sided [5.84 to 50.46] — Difference in Least Squares Means (back-transformation of difference in log-fractions from baseline)

11. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Serum Bone-specific Alkaline Phosphatase [s-BSAP]) at 12 Months
Description: Back-transformation (geometric mean) of the Least Squares Mean of the log-values Percentage change from baseline, in Biochemical Marker of Bone turnover (serum bone-specific alkaline phosphatase (s-BSAP)), at 12 Months
Time Frame: Baseline and 12 months
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base
Number analyzed (Participants) | 62 | 58 | 57 | 64 | 58
Percentage change | -2.77 [-10.39 to 5.49] | 42.08 [30.64 to 54.52] | 8.95 [0.10 to 18.60] | 2.66 [-5.25 to 11.24] | -18.35 [-24.93 to -11.18]
Statistical Analysis 1: Comparison: Placebo-Base vs Odanacatib 50 Mg-Base; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on biochemical indices of bone formation (s-BSAP) compared to placebo over 12 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -15.57, 95% CI 2-sided [-26.11 to -5.04] — Difference in Least Squares Means (back-transformation from difference in log-fraction from baseline)
Statistical Analysis 2: Comparison: Placebo-Base vs Odanacatib 25 Mg-Base; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.645, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = 5.43, 95% CI 2-sided [-6.02 to 16.89] — Difference in Least Squares Means (back-transformation from difference in log-fraction from baseline)
Statistical Analysis 3: Comparison: Placebo-Base vs Odanacatib 10 Mg-Base; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; ANCOVA — Significance for secondary endpoints was only declared if there was also significance for the primary endpoint. Multiplicity was addressed through stepdown trend-test approach. Multiplicity for multiple endpoints was handle by a Hochberg procedure; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = 11.73, 95% CI 2-sided [-0.47 to 23.92] — Difference in Least Squares Means (back-transformation from difference in log-fraction from baseline)
Statistical Analysis 4: Comparison: Placebo-Base vs Odanacatib 3 Mg-Base; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = 44.85, 95% CI 2-sided [30.55 to 59.16] — Difference in Least Squares Means (back-transformation from difference in log-fraction from baseline)

12. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Serum N-Terminal Propeptide of Type 1 Collagen [s-P1NP]) at 12 Months
Description: Back-transformation (geometric mean) of the Least Squares Mean of the log-values Percentage change in Biochemical Marker of Bone turnover (serum N-terminal propeptide of Type 1 collagen (s-P1NP) (relative to baseline) at 12 Months
Time Frame: Baseline and 12 months
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Base | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base
Number analyzed (Participants) | 62 | 57 | 57 | 63 | 58
Percentage change | 3.91 [-8.79 to 18.38] | 50.81 [31.69 to 72.70] | 2.33 [-10.63 to 17.16] | 2.23 [-10.12 to 16.28] | -31.83 [-40.40 to -22.02]
Statistical Analysis 1: Comparison: Placebo-Base vs Odanacatib 50 Mg-Base; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on biochemical indices of bone formation (s-P1NP) compared to placebo over 12 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -35.74, 95% CI 2-sided [-52.14 to -19.33] — Difference in Least Squares Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 2: Comparison: Placebo-Base vs Odanacatib 25 Mg-Base; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.161, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -1.68, 95% CI 2-sided [-20.58 to 17.23] — Difference in Least Squares Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 3: Comparison: Placebo-Base vs Odanacatib 10 Mg-Base; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 11, analysis 3]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -1.58, 95% CI 2-sided [-20.99 to 17.82] — Difference in Least Squares Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 4: Comparison: Placebo-Base vs Odanacatib 3 Mg-Base; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 11, analysis 3]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = 46.90, 95% CI 2-sided [22.35 to 71.44] — Difference in Least Squares Means (back-transformation of difference in log-fraction from baseline)

13. Secondary Outcome: Percentage Change From Baseline in Total Hip Bone Mineral Density at 24 Months
Description: Percentage change in total hip Bone Mineral Density (relative to baseline) at 24 Months
Time Frame: Baseline and 24 months
Population: This analysis was performed at Month 24 using Full-Analysis-Set Population with Last Observation Carried Forward (from extension data). No data was carried forward from the core to the extension period.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1
Number analyzed (Participants) | 61 | 57 | 59 | 65 | 58
Percentage change | -0.93 [-1.86 to -0.01] | -1.44 [-2.40 to -0.48] | 1.82 [0.88 to 2.76] | 2.55 [1.66 to 3.44] | 3.16 [2.22 to 4.11]
Statistical Analysis 1: Comparison: Placebo-Ext 1 vs Odanacatib 50 Mg-Ext 1; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on total hip BMD compared to placebo over 24 months. The secondary hypothesis states that odanacatib will increase total hip BMD compared to placebo over 24 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 4.10, 95% CI 2-sided [2.77 to 5.42]
Statistical Analysis 2: Comparison: Placebo-Ext 1 vs Odanacatib 25 Mg-Ext 1; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 3.48, 95% CI 2-sided [2.20 to 4.77]
Statistical Analysis 3: Comparison: Placebo-Ext 1 vs Odanacatib 10 Mg-Ext 1; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 2.75, 95% CI 2-sided [1.43 to 4.07]
Statistical Analysis 4: Comparison: Placebo-Ext 1 vs Odanacatib 3 Mg-Ext 1; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.536, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.51, 95% CI 2-sided [-1.84 to 0.83]

14. Secondary Outcome: Percentage Change From Baseline in Femoral Neck BMD at 24 Months
Description: Percentage change in femoral neck Bone Mineral Density (relative to baseline) at 24 Months
Time Frame: Baseline and 24 months
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1
Number analyzed (Participants) | 61 | 57 | 59 | 65 | 58
Percentage change | -0.85 [-1.85 to 0.16] | -1.25 [-2.29 to -0.22] | 1.97 [0.95 to 2.98] | 2.73 [1.76 to 3.69] | 3.84 [2.82 to 4.86]
Statistical Analysis 1: Comparison: Placebo-Ext 1 vs Odanacatib 50 Mg-Ext 1; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on femoral neck BMD compared to placebo over 24 months. The secondary hypothesis states that odanacatib will increase femoral neck BMD compared to placebo over 24 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 4.69, 95% CI 2-sided [3.25 to 6.12]
Statistical Analysis 2: Comparison: Placebo-Ext 1 vs Odanacatib 25 Mg-Ext 1; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Square Means = 3.57, 95% CI 2-sided [2.18 to 4.97]
Statistical Analysis 3: Comparison: Placebo-Ext 1 vs Odanacatib 10 Mg-Ext 1; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 2.82, 95% CI 2-sided [1.39 to 4.25]
Statistical Analysis 4: Comparison: Placebo-Ext 1 vs Odanacatib 3 Mg-Ext 1; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.585, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.41, 95% CI 2-sided [-1.85 to 1.04]

15. Secondary Outcome: Percentage Change From Baseline in Trochanter BMD at 24 Months
Description: Percentage change from baseline in trochanter BMD (relative to baseline) at 24 Months
Time Frame: Baseline and 24 months
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1
Number analyzed (Participants) | 61 | 57 | 59 | 65 | 58
Percentage Change | -0.81 [-2.15 to 0.53] | -0.85 [-2.23 to 0.53] | 3.61 [2.26 to 4.97] | 3.75 [2.46 to 5.04] | 4.28 [2.92 to 5.65]
Statistical Analysis 1: Comparison: Placebo-Ext 1 vs Odanacatib 50 Mg-Ext 1; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on trochanter BMD compared to placebo over 24 months. The secondary hypothesis states that odanacatib will increase trochanter BMD compared to placebo over 24 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 5.09, 95% CI 2-sided [3.18 to 7.01]
Statistical Analysis 2: Comparison: Placebo-Ext 1 vs Odanacatib 25 Mg-Ext 1; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 4.56, 95% CI 2-sided [2.70 to 6.42]
Statistical Analysis 3: Comparison: Placebo-Ext 1 vs Odanacatib 10 Mg-Ext 1; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = 4.43, 95% CI 2-sided [2.52 to 6.33]
Statistical Analysis 4: Comparison: Placebo-Ext 1 vs Odanacatib 3 Mg-Ext 1; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.981, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -0.04, 95% CI 2-sided [-1.97 to 1.89]

16. Secondary Outcome: Percentage Change From Baseline in Total Body BMD at 24 Months
Description: Percentage change in total body BMD (relative to baseline) at 24 Months
Time Frame: Baseline and 24 months
Population: This analysis was performed at Month 24 using Full-Analysis-Set Population with Last Observation Carried Forward. No data was carried forward from the core to the extension period.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1
Number analyzed (Participants) | 56 | 47 | 48 | 58 | 51
Percentage change | -1.54 [-2.42 to -0.66] | -2.70 [-3.66 to -1.74] | -1.35 [-2.29 to -0.40] | -0.43 [-1.29 to 0.43] | 0.19 [-0.73 to 1.11]
Statistical Analysis 1: Comparison: Placebo-Ext 1 vs Odanacatib 50 Mg-Ext 1; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on Total Body BMD compared to placebo over 24 months. The secondary hypothesis states that odanacatib will increase Total Body BMD compared to placebo over 24 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least square means = 1.73, 95% CI [0.46 to 3.01]
Statistical Analysis 2: Comparison: Placebo-Ext 1 vs Odanacatib 25 Mg-Ext 1; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.028, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least square means = 1.11, 95% CI [-0.12 to 2.34]
Statistical Analysis 3: Comparison: Placebo-Ext 1 vs Odanacatib 10 Mg-Ext 1; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p = 0.804, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in Least square means = 0.20, 95% CI [-1.10 to 1.49]
Statistical Analysis 4: Comparison: Placebo-Ext 1 vs Odanacatib 3 Mg-Ext 1; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least square means = -1.15, 95% CI 2-sided [-2.46 to 0.15]

17. Secondary Outcome: Percentage Change From Baseline in Distal Forearm BMD at 24 Months
Description: Percentage change in distal forearm BMD (relative to baseline) at 24 Months
Time Frame: Baseline and 24 months
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base
Number analyzed (Participants) | 61 | 58 | 60 | 65 | 57
Percentage change | -2.75 [-3.83 to -1.66] | -5.70 [-6.80 to -4.59] | -1.22 [-2.31 to -0.13] | -0.65 [-1.70 to 0.39] | 0.15 [-0.97 to 1.27]
Statistical Analysis 1: Comparison: Placebo-Base vs Odanacatib 50 Mg-Base; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on Distal Forearm BMD compared to placebo over 24 months. The secondary hypothesis states that odanacatib will increase Distal Forearm BMD compared to placebo over 24 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least square means = 2.90, 95% CI 2-sided [1.34 to 4.46]
Statistical Analysis 2: Comparison: Placebo-Base vs Odanacatib 25 Mg-Base; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least square means = 2.09, 95% CI [0.59 to 3.60]
Statistical Analysis 3: Comparison: Placebo-Base vs Odanacatib 10 Mg-Ext 1; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.094, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 1, analysis 1]; Difference in Least square means = 1.53, 95% CI [-0.01 to 3.07]
Statistical Analysis 4: Comparison: Placebo-Base vs Odanacatib 3 Mg-Base; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; ANCOVA — [p-value comment as in outcome 11, analysis 3]; [statistical method as in outcome 1, analysis 1]; Difference in Least square means = -2.95, 95% CI [-4.50 to -1.40]

18. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Urinary N-Telopeptides of Type I Collagen [u-NTx]) at 24 Months
Description: Back-transformation (geometric mean) of the Least Squares Mean of the log-values percentage change from baseline in biochemical marker of bone turnover (u-NTx) (relative to baseline) at 24 Months
Time Frame: Baseline and 24 months
Population: Analysis used a geometric mean percent change from baseline (back-transformation of a log-transformed fraction from baseline) at Month 24 using a Per-Protocol approach. Participants with important protocol deviations and major protocol violators were excluded from the analyses. The Per-Protocol approach did not estimate missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Base | Odanacatib 3 Mg-Base | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Base | Odanacatib 50 Mg-Base
Number analyzed (Participants) | 56 | 45 | 41 | 51 | 38
Percentage change | -4.62 [-18.23 to 11.25] | 12.89 [-4.93 to 34.05] | -40.57 [-50.32 to -28.90] | -38.30 [-47.48 to -27.51] | -51.83 [-60.05 to -41.91]
Statistical Analysis 1: Comparison: Placebo-Base vs Odanacatib 50 Mg-Base; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on biochemical indices of bone resorption (u-NTx) compared to placebo over 24 months. The secondary hypothesis states that odanacatib will decrease biochemical indices of bone resorption (u-NTx) over 24 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = -47.21, 95% CI [-64.51 to -29.90] — Difference in Least Square Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 2: Comparison: Placebo-Base vs Odanacatib 25 Mg-Base; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = -33.67, 95% CI [-51.44 to -15.91] — Difference in Least Square Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 3: Comparison: Placebo-Base vs Odanacatib 10 Mg-Ext 1; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = -35.94, 95% CI [-54.15 to -17.74] — Difference in Least Square Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 4: Comparison: Placebo-Base vs Odanacatib 3 Mg-Base; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.101, ANCOVA — [p-value comment as in outcome 11, analysis 3]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = 17.51, 95% CI 2-sided [-6.78 to 41.80] — Difference in Least Square Means (back-transformation of difference in log-fraction from baseline)

19. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Serum C-Telopeptides of Type 1 Collagen [s-CTx]) at 24 Months
Description: Back-transformation (geometric mean) of the Least Squares Mean of the log-values Percentage change from baseline, in Biochemical Marker of Bone turnover (serum C-telopeptides of Type 1 collagen (s-CTx)) (relative to baseline) at 24 Months
Time Frame: Baseline and 24 months
Population: Analysis used geometric mean percent change from baseline (back-transformation of a log-transformed fraction from baseline) at Month 24 using a Per-Protocol approach. Participants with important protocol deviations and major protocol violators were excluded from the analyses. The per-protocol approach did not estimate missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1
Number analyzed (Participants) | 56 | 45 | 42 | 52 | 39
Percentage change | 32.77 [13.28 to 55.61] | 54.94 [29.83 to 84.92] | 8.79 [-9.35 to 30.57] | -6.52 [-20.70 to 10.19] | -30.57 [-42.60 to -16.20]
Statistical Analysis 1: Comparison: Placebo-Ext 1 vs Odanacatib 50 Mg-Ext 1; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on biochemical indices of bone resorption (s-CTx) compared to placebo over 24 months. The secondary hypothesis states that odanacatib will decrease biochemical indices of bone resorption (s-CTx) over 24 months; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = -63.34, 95% CI [-88.32 to -38.36] — Difference in Least Square Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 2: Comparison: Placebo-Ext 1 vs Odanacatib 25 Mg-Ext 1; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p <= 0.001, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -39.29, 95% CI 2-sided [-65.40 to -13.18] — Difference in Least Squares Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 3: Comparison: Placebo-Ext 1 vs Odanacatib 10 Mg-Ext 1; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.124, ANCOVA — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -23.98, 95% CI 2-sided [-53.04 to 5.09] — Difference in Least Squares Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 4: Comparison: Placebo-Ext 1 vs Odanacatib 3 Mg-Ext 1; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = 22.18, 95% CI 2-sided [-12.38 to 56.73] — Difference in Least Squares Means (back-transformation of difference in log-fraction from baseline)

20. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Urinary Total Deoxypyridinolines [u-DPyr]) at 24 Months
Description: Back-transformation (geometric mean) of the Least Squares Mean of the log-values Percentage change from baseline, in Biochemical Marker of Bone turnover (urinary total deoxypyridinolines (u-DPyr)) (relative to baseline) at 24 Months
Time Frame: Baseline and 24 months
Population: as for outcome 19
Measure: Least Squares Mean (95% Confidence Interval); unit: Geometric LS Mean percent change
Arm/Group | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1
Number analyzed (Participants) | 56 | 45 | 40 | 51 | 38
Geometric LS Mean percent change | -5.78 [-18.44 to 8.84] | 15.96 [-1.29 to 36.23] | -7.57 [-22.03 to 9.57] | -14.30 [-26.30 to -0.33] | -22.49 [-34.96 to -7.64]
Statistical Analysis 1: Comparison: Placebo-Ext 1 vs Odanacatib 50 Mg-Ext 1; The secondary objective was to assess the effect of MK0822 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on biochemical indices of bone resorption (u-DPyr) compared to placebo over 24 months. The secondary hypothesis states that MK0822 will decrease biochemical indices of bone resorption (u-DPyr) over 24 months; Test type: Superiority or Other; p = 0.015, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = -16.71, 95% CI [-36.03 to 2.61] — Difference in Least Square Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 2: Comparison: Placebo-Ext 1 vs Odanacatib 25 Mg-Ext 1; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.246, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = -8.51, 95% CI [-27.31 to 10.29] — Difference in Least Square Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 3: Comparison: Placebo-Ext 1 vs Odanacatib 10 Mg-Ext 1; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = -1.79, 95% CI [-22.66 to 19.08] — Difference in Least Square Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 4: Comparison: Placebo-Ext 1 vs Odanacatib 3 Mg-Ext 1; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = 21.74, 95% CI [-1.32 to 44.81] — Difference in Least Square Means (back-transformation of difference in log-fraction from baseline)

21. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Serum Bone-specific Alkaline Phosphatase [s-BSAP]) at 24 Months
Description: Back-transformation (geometric mean) of the Least Squares Mean of the log-values Percentage change from baseline, in Biochemical Marker of Bone turnover (serum bone-specific alkaline phosphatase (s-BSAP)) (relative to baseline) at 24 Months
Time Frame: Baseline and 24 months
Population: as for outcome 19
Measure: Least Squares Mean (95% Confidence Interval); unit: Geometric LS Mean percent change
Arm/Group | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1
Number analyzed (Participants) | 57 | 47 | 42 | 53 | 42
Geometric LS Mean percent change | 3.38 [-4.94 to 12.44] | 40.17 [27.80 to 53.73] | 2.99 [-6.57 to 13.54] | 10.62 [1.40 to 20.69] | -13.62 [-21.36 to -4.32]
Statistical Analysis 1: Comparison: Placebo-Ext 1 vs Odanacatib 50 Mg-Ext 1; The secondary objective was to assess the effect of MK0822 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on biochemical indices of bone formation (s-BSAP) compared to placebo over 24 months; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = -16.64, 95% CI [-28.84 to -4.44] — Difference in Least Square Means (back-transformation of difference in log-fractions from baseline)
Statistical Analysis 2: Comparison: Placebo-Ext 1 vs Odanacatib 25 Mg-Ext 1; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.852, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = 7.24, 95% CI [-5.73 to 20.21] — Difference in Least Square Means (back-transformation of difference in log-fractions from baseline)
Statistical Analysis 3: Comparison: Placebo-Ext 1 vs Odanacatib 10 Mg-Ext 1; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = -0.39, 95% CI [-13.69 to 12.92] — Difference in Least Square Means (back-transformation of difference in log-fractions from baseline)
Statistical Analysis 4: Comparison: Placebo-Ext 1 vs Odanacatib 3 Mg-Ext 1; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = 36.79, 95% CI [21.19 to 52.38] — Difference in Least Square Means (back-transformation of difference in log-fractions from baseline)

22. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Serum N-Terminal Propeptide of Type 1 Collagen [s-P1NP]) at 24 Months
Description: Back-transformation (geometric mean) of the least squares mean of the log-values percentage change from baseline in biochemical marker of bone turnover (s-P1NP) (relative to baseline) at 24 months
Time Frame: Baseline and 24 months
Population: as for outcome 19
Measure: Least Squares Mean (95% Confidence Interval); unit: Geometric LS Mean percent change
Arm/Group | Placebo-Ext 1 | Odanacatib 3 Mg-Ext 1 | Odanacatib 10 Mg-Ext 1 | Odanacatib 25 Mg-Ext 1 | Odanacatib 50 Mg-Ext 1
Number analyzed (Participants) | 57 | 47 | 42 | 53 | 42
Geometric LS Mean percent change | 1.29 [-11.11 to 15.43] | 50.52 [30.37 to 73.79] | 9.07 [-6.28 to 26.93] | 14.60 [0.08 to 31.23] | -20.20 [-31.49 to -7.05]
Statistical Analysis 1: Comparison: Placebo-Ext 1 vs Odanacatib 50 Mg-Ext 1; The secondary objective was to assess the effect of odanacatib 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on biochemical indices of bone formation (s-P1NP) compared to placebo over 24 months; Test type: Superiority or Other; p = 0.011, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 8, analysis 1]; Difference in Least Squares Means = -21.49, 95% CI 2-sided [-39.55 to -3.43] — Difference in Least Squares Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 2: Comparison: Placebo-Ext 1 vs Odanacatib 25 Mg-Ext 1; The secondary objective was to assess the effect of MK0822 3 mg weekly, 10 mg weekly, 25 mg weekly, and 50 mg weekly on biochemical indices of bone formation (s-P1NP) compared to placebo over 24 months; Test type: Superiority or Other; p = 0.618, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 8, analysis 1]; Difference in Least square means = 13.31, 95% CI [-7.10 to 33.71] — Difference in Least square means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 3: Comparison: Placebo-Ext 1 vs Odanacatib 10 Mg-Ext 1; [analysis description as in outcome 22, analysis 1]; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 8, analysis 1]; Difference in Least square means = 7.77, 95% CI 2-sided [-13.46 to 29.01] — Difference in Least Squares Means (back-transformation of difference in log-fraction from baseline)
Statistical Analysis 4: Comparison: Placebo-Ext 1 vs Odanacatib 3 Mg-Ext 1; [analysis description as in outcome 22, analysis 1]; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 8, analysis 1]; Difference in Least Square Means = 49.23, 95% CI 2-sided [23.86 to 74.59] — Difference in Least Square Means (back-transformation of difference in log-fraction from baseline)

23. Primary Outcome: Percentage Change From Baseline in Lumbar Spine BMD at 36 Months
Description: Percentage change in lumbar spine BMD (relative to baseline) at 36 months
Time Frame: Baseline and 36 months
Population: This analysis was performed at Month 36 using the Per-protocol approach which includes patients who took at least one dose of extension study medication and had the necessary follow-up information. Missing values were not imputed. No data were carried forward from month 30 to 36.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Groups:
- Odanacatib 25 mg / 50 Mg-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one placebo tablet once a week. Before entering this extension, participants in this treatment group had taken one 25 mg tablet of odanacatib once a week for 2 years.
Arm/Group | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / Placebo-Ext 2 | Odanacatib 25 mg / 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2
Number analyzed (Participants) | 14 | 16 | 17 | 13 | 12 | 10 | 12 | 18 | 15 | 17
Percent Change | 0.42 [-1.89 to 2.73] | 2.95 [0.79 to 5.11] | -1.57 [-3.67 to 0.54] | 4.41 [2.01 to 6.82] | 2.03 [-0.47 to 4.53] | 6.11 [3.37 to 8.85] | 0.32 [-2.18 to 2.82] | 7.45 [5.41 to 9.48] | 1.39 [-0.84 to 3.63] | 7.85 [5.74 to 9.95]
Statistical Analysis 1: Comparison: Odanacatib 50 mg / Placebo-Ext 2 vs Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2; In postmenopausal women with osteoporosis assess the time course of resolution of effect on lumbar spine BMD during the 12 month extension following 24 months of treatment with odanacatib once weekly. The primary objective was to assess the resolution of effect, on lumbar spine BMD, for the participants who received odanacatib 50 mg for 3 years compared to those who received odanacatib 50 mg in the 2nd year and switched to placebo for the 3rd year extension; Test type: Superiority or Other; Difference in Least Square Means = 6.45, 95% CI 2-sided [3.38 to 9.53]

24. Secondary Outcome: Percentage Change From Baseline in Total Hip BMD at 36 Months
Description: Percentage change in total hip BMD (relative to baseline) at 36 months
Time Frame: Baseline and 36 months
Population: This analysis was performed at Month 36 using the Per-Protocol approach which includes participants who took at least one dose of extension study medication and had the necessary follow-up information. Missing values were not imputed. No data were carried forward from month 30 to 36.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / 50 Mg-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2
Number analyzed (Participants) | 14 | 16 | 17 | 12 | 11 | 9 | 12 | 19 | 15 | 17
Percentage change | -0.77 [-2.92 to 1.38] | 1.16 [-0.86 to 3.17] | -0.63 [-2.59 to 1.33] | 2.75 [0.42 to 5.07] | 0.96 [-1.48 to 3.39] | 4.61 [1.93 to 7.30] | 1.64 [-0.69 to 3.97] | 5.70 [3.85 to 7.54] | -0.48 [-2.56 to 1.60] | 5.83 [3.87 to 7.79]
Statistical Analysis 1: Comparison: Odanacatib 50 mg / Placebo-Ext 2 vs Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2; Test type: Superiority or Other; Difference in Least Square Means = 6.31, 95% CI 2-sided [3.44 to 9.17]

25. Secondary Outcome: Percentage Change From Baseline in Femoral Neck BMD at 36 Months
Description: Percentage change in femoral neck BMD (relative to baseline) at 36 Months
Time Frame: Baseline and 36 months
Population: as for outcome 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / 50 Mg-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2
Number analyzed (Participants) | 14 | 16 | 17 | 12 | 11 | 9 | 12 | 19 | 15 | 17
Percentage change | -0.52 [-2.67 to 1.63] | 1.03 [-0.98 to 3.04] | -1.04 [-2.99 to 0.92] | 2.26 [-0.06 to 4.59] | -0.14 [-2.57 to 2.30] | 5.06 [2.38 to 7.74] | 0.80 [-1.52 to 3.13] | 7.23 [5.38 to 9.07] | 2.26 [0.19 to 4.34] | 4.97 [3.01 to 6.93]
Statistical Analysis 1: Comparison: Odanacatib 50 mg / Placebo-Ext 2 vs Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2; Test type: Superiority or Other; Difference in Least Square Means = 2.71, 95% CI 2-sided [-0.16 to 5.57]

26. Secondary Outcome: Percentage Change From Baseline in Trochanter BMD at 36 Months
Description: Percentage change in trochanter BMD (relative to baseline) at 36 months
Time Frame: Baseline and 36 months
Population: as for outcome 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / 50 Mg-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2
Number analyzed (Participants) | 14 | 16 | 17 | 12 | 11 | 9 | 12 | 19 | 15 | 17
Percentage Change | -0.46 [-3.71 to 2.79] | 2.32 [-0.72 to 5.36] | -1.04 [-4.00 to 1.92] | 4.53 [1.01 to 8.04] | 0.66 [-3.02 to 4.34] | 8.21 [4.16 to 12.27] | 1.14 [-2.38 to 4.65] | 7.97 [5.18 to 10.76] | -0.69 [-3.83 to 2.46] | 7.44 [4.48 to 10.41]
Statistical Analysis 1: Comparison: Odanacatib 50 mg / Placebo-Ext 2 vs Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2; Test type: Superiority or Other; Difference in Least Square Means = 8.13, 95% CI 2-sided [3.80 to 12.46]

27. Secondary Outcome: Percentage Change From Baseline in Total Body BMD at 36 Months
Description: Percentage change from baseline in total body BMD (relative to baseline) at 36 Months
Time Frame: Baseline and 36 months
Population: as for outcome 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / 50 Mg-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2
Number analyzed (Participants) | 14 | 14 | 16 | 13 | 12 | 9 | 12 | 18 | 15 | 17
Percentage change | 0.13 [-2.12 to 2.38] | -2.20 [-4.45 to 0.05] | -3.63 [-5.74 to -1.52] | 0.28 [-2.07 to 2.62] | -2.28 [-4.71 to 0.15] | -1.22 [-4.03 to 1.58] | -0.85 [-3.29 to 1.58] | 0.56 [-1.43 to 2.54] | -1.84 [-4.02 to 0.34] | -0.38 [-2.43 to 1.67]
Statistical Analysis 1: Comparison: Odanacatib 50 mg / Placebo-Ext 2 vs Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2; Test type: Superiority or Other; Difference in Least Square Means = 1.46, 95% CI 2-sided [-1.54 to 4.46]

28. Secondary Outcome: Percentage Change From Baseline in Distal Forearm BMD at 36 Months
Description: Percentage change in distal forearm BMD (relative to baseline) at 36 Months
Time Frame: Baseline and 36 months
Population: as for outcome 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / 50 Mg-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2
Number analyzed (Participants) | 14 | 15 | 16 | 13 | 12 | 10 | 12 | 18 | 14 | 17
Percentage Change | -2.08 [-4.60 to 0.43] | -4.04 [-6.47 to -1.61] | -6.59 [-8.95 to -4.23] | -6.34 [-8.96 to -3.73] | -1.74 [-4.46 to 0.97] | -3.74 [-6.71 to -0.76] | -2.39 [-5.11 to 0.32] | 0.53 [-1.69 to 2.74] | -2.73 [-5.25 to -0.22] | -0.26 [-2.55 to 2.03]
Statistical Analysis 1: Comparison: Odanacatib 50 mg / Placebo-Ext 2 vs Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2; Test type: Superiority or Other; Difference in Least Square Means = 2.47, 95% CI 2-sided [-0.93 to 5.88]

29. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Urinary N-Telopeptides of Type I Collagen [u-NTx]) at 36 Months
Description: Percentage change from baseline in biochemical marker of bone turnover (u-NTx) at 36 Months
Time Frame: Baseline and 36 months
Population: This analysis was geometric mean percent change from baseline (which is a back-transformation of a log-transformed fraction from baseline) at Month 36 using a Per-Protocol approach. Participants with important protocol deviations and major protocol violators were excluded from the analyses. The Per-Protocol approach did not estimate missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / 50 Mg-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2
Number analyzed (Participants) | 14 | 15 | 13 | 16 | 13 | 11 | 10 | 18 | 14 | 17
Percentage change | -17.43 [-39.06 to 11.86] | -55.12 [-66.51 to 39.85] | -11.90 [-35.76 to 20.83] | -57.17 [-67.75 to -43.12] | -12.15 [-35.91 to 20.43] | -49.10 [-63.88 to -28.27] | 14.26 [-20.17 to 63.53] | -52.11 [-63.33 to -37.45] | 27.55 [-5.86 to 72.80] | -50.51 [-62.44 to -34.81]
Statistical Analysis 1: Comparison: Odanacatib 50 mg / Placebo-Ext 2 vs Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2; Test type: Superiority or Other; Difference in Least Square Means = -78.06, 95% CI 2-sided [-119.20 to -36.92]

30. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Serum C-Telopeptides of Type 1 Collagen [s-CTx]) at 36 Months
Description: Percentage change from baseline in biochemical marker of bone turnover (s-CTx) at 36 Months
Time Frame: Baseline and 36 months
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / 50 Mg-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2
Number analyzed (Participants) | 14 | 15 | 13 | 16 | 13 | 11 | 9 | 18 | 14 | 17
Percentage change | -0.09 [-28.93 to 40.46] | -41.30 [-57.74 to -18.47] | -4.69 [-33.13 to 35.85] | -44.62 [-59.72 to -23.88] | 18.24 [-16.98 to 68.41] | -26.26 [-49.81 to 8.33] | 61.14 [5.50 to 146.12] | -36.71 [-53.09 to -14.60] | 10.32 [-21.52 to 55.10] | -23.93 [-44.15 to 3.63]
Statistical Analysis 1: Comparison: Odanacatib 50 mg / Placebo-Ext 2 vs Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2; Test type: Superiority or Other; Difference in Least Square Means = -34.25, 95% CI 2-sided [-78.70 to 10.20]

31. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Urinary Total Deoxypyridinolines [u-DPyr]) at 36 Months
Description: Percentage change from baseline in biochemical marker of bone turnover u-DPyr at 36 Months
Time Frame: Baseline and 36 months
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / 50 Mg-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2
Number analyzed (Participants) | 14 | 15 | 13 | 14 | 13 | 11 | 10 | 18 | 14 | 17
Percentage change | -18.69 [-41.68 to 13.36] | -14.95 [-38.27 to 17.18] | -7.82 [-34.76 to 30.26] | -26.27 [-47.10 to 2.76] | -4.69 [-32.51 to 34.60] | 0.43 [-31.00 to 46.19] | -9.16 [-38.64 to 34.48] | -16.41 [-37.59 to 11.97] | 22.41 [-12.20 to 70.66] | -16.84 [-38.49 to 12.45]
Statistical Analysis 1: Comparison: Odanacatib 50 mg / Placebo-Ext 2 vs Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2; Test type: Superiority or Other; Difference in Least Square Means = -39.25, 95% CI 2-sided [-87.17 to 8.68]

32. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Serum Bone-specific Alkaline Phosphatase [s-BSAP]) at 36 Months
Description: Geometric Mean Percentage change from baseline, in Biochemical Marker of Bone turnover (serum bone-specific alkaline phosphatase [s-BSAP]) at 36 Months
Time Frame: Baseline and 36 months
Population: This analysis was geometric mean percent change from baseline (which is a back-transformation of a log-transformed fraction from baseline) at Month 36 using a Per-Protocol approach where patients with important protocol deviations and major protocol violators were excluded from the analyses. The per-protocol approach did not estimate missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Geometric Mean Percent Change
Arm/Group | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / 50 Mg-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2
Number analyzed (Participants) | 14 | 16 | 14 | 16 | 13 | 11 | 12 | 18 | 14 | 17
Geometric Mean Percent Change | 7.73 [-7.32 to 25.24] | 10.86 [-3.69 to 27.62] | 14.26 [-1.77 to 32.91] | 9.13 [-5.20 to 25.62] | 12.95 [-3.41 to 32.08] | 8.49 [-8.48 to 28.62] | 33.74 [13.71 to 57.31] | 11.12 [-2.67 to 26.86] | 1.30 [-12.85 to 17.76] | 17.90 [2.83 to 35.17]
Statistical Analysis 1: Comparison: Odanacatib 50 mg / Placebo-Ext 2 vs Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2; Test type: Superiority or Other; Difference in Least Square Means = 16.59, 95% CI 2-sided [-5.67 to 38.85]

33. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Serum N-terminal Propeptide of Type 1 Collagen [s-P1NP]) at 36 Months
Description: Percentage change from baseline in biochemical marker of bone turnover (serum N-terminal propeptide of Type 1 collagen [s-P1NP]) at 36 months
Time Frame: Baseline and 36 months
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / 50 Mg-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2
Number analyzed (Participants) | 14 | 16 | 14 | 15 | 13 | 11 | 12 | 18 | 14 | 17
Percentage change | -20.79 [-40.08 to 4.72] | -18.79 [-37.44 to 5.42] | -13.11 [-34.35 to 15.00] | -21.08 [-39.75 to 3.37] | 8.58 [-18.75 to 45.11] | 12.44 [-17.98 to 54.13] | 22.57 [-9.27 to 65.59] | -8.14 [-28.14 to 17.42] | -0.77 [-24.94 to 31.18] | -6.20 [-27.20 to 20.86]
Statistical Analysis 1: Comparison: Odanacatib 50 mg / Placebo-Ext 2 vs Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2; Test type: Superiority or Other; Difference in Least Square Means = -5.43, 95% CI 2-sided [-42.04 to 31.18]

34. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Serum Bone Tartrate-resistant Acid Phosphatase Isoform 5b [TRAP 5-b]) at 36 Months
Description: Percentage change from baseline in biochemical marker of bone turnover (serum bone tartrate-resistant acid phosphatase isoform 5b [TRAP 5-b]) at 36 Months
Time Frame: Baseline and 36 months
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / 50 Mg-Ext 2 | Odanacatib 25 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2
Number analyzed (Participants) | 10 | 11 | 10 | 12 | 10 | 9 | 10 | 15 | 10 | 15
Percentage change | 52.98 [29.87 to 80.21] | 52.37 [30.34 to 78.12] | 33.25 [13.12 to 56.97] | 59.37 [37.24 to 85.08] | 56.71 [33.04 to 84.60] | 82.94 [53.93 to 117.42] | 56.42 [32.79 to 84.26] | 77.90 [55.63 to 103.36] | 47.61 [25.30 to 73.88] | 96.70 [72.08 to 124.85]
Statistical Analysis 1: Comparison: Odanacatib 50 mg / Placebo-Ext 2 vs Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2; Test type: Superiority or Other; Difference in Least Square Means = 49.10, 95% CI 2-sided [13.37 to 84.83]

35. Secondary Outcome: Percentage Change From Baseline in Biochemical Marker of Bone Turnover (Serum Cross-Linked Carboxyterminal Telopeptides of Type I Collagen [1-CTP]) at 36 Months
Description: Percentage change from baseline in biochemical marker of bone turnover (serum Cross-Linked Carboxyterminal Telopeptides of Type I Collagen [1-CTP]) at 36 Months
Time Frame: Baseline and 36 months
Population: as for outcome 29
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Groups:
- Odanacatib 25 mg / Placebo 50 Mg-Ext 2: 12 Month Extension (Year 3)
  During this 12 month extension patients in this treatment group took one placebo tablet once a week. Patients in this treatment group took one 25 mg tablet of MK0822 once a week during 2 years and one placebo tablet once a week during the 3rd year.
Arm/Group | Placebo / Placebo-Ext 2 | Placebo / Odanacatib 50 Mg-Ext 2 | Odanacatib 3 mg / Placebo-Ext 2 | Odanacatib 3 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 10 mg / Placebo-Ext 2 | Odanacatib 10 mg / Odanacatib 50 Mg-Ext 2 | Odanacatib 25 mg / Placebo 50 Mg-Ext 2 | Odanacatib 25 mg / 50 Mg-Ext 2 | Odanacatib 50 mg / Placebo-Ext 2 | Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2
Number analyzed (Participants) | 14 | 13 | 14 | 16 | 12 | 11 | 11 | 19 | 15 | 18
Percentage change | 7.40 [-16.78 to 38.60] | 193.91 [125.61 to 282.89] | 1.67 [-21.41 to 31.53] | 187.37 [126.25 to 264.99] | 58.76 [20.27 to 109.56] | 188.50 [116.34 to 284.74] | 77.94 [33.46 to 137.24] | 231.93 [166.74 to 313.05] | 27.20 [-0.61 to 62.79] | 236.64 [168.69 to 321.76]
Statistical Analysis 1: Comparison: Odanacatib 50 mg / Placebo-Ext 2 vs Odanacatib 50 mg / Odanacatib 50 Mg-Ext 2; Test type: Superiority or Other; Difference in Least Squares Means = 209.44, 95% CI 2-sided [127.14 to 291.73]

36. Primary Outcome: Percentage Change From Baseline in Lumbar Spine BMD at 60 Months
Description: Percentage change from baseline in lumbar spine BMD at 60 months.
Time Frame: Baseline and Month 60
Population: All participants who took at least one dose of base study medication and at least one dose of extension medication. Missing values were imputed using last observation-carried-forward principle.
Measure: Mean (95% Confidence Interval); unit: Percentage change
Groups:
- Placebo Once Weekly: One placebo tablet once a week
- Odanacatib 50 mg Once Weekly: One odanacatib 50 mg tablet once a week
Arm/Group | Placebo Once Weekly | Odanacatib 50 mg Once Weekly
Number analyzed (Participants) | 14 | 13
Percentage change | -0.41 [-3.1 to 2.28] | 11.88 [7.23 to 16.54]

37. Primary Outcome: Percentage Change From Baseline in Lumbar Spine BMD at 120 Months
Description: Percentage change from baseline in lumbar spine BMD at 120 Months.
Time Frame: Baseline and Month 120
Population: This analysis was based on the FAS population, which included all randomized participants who took at least 1 dose of extension study drug and had the necessary extension data available for this endpoint. Missing data were not imputed.
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Groups:
- Group A: Odanacatib 50 mg Once Weekly: Group A consists of a combination of participants who were treated with odanacatib 25 mg for 2 years, then odanacatib 50 mg for 8 years; and participants who were treated with odanacatib 50 mg for 10 years.
- Group B: Odanacatib 50 mg Once Weekly: Group B consists of a combination participants who were treated with placebo for 2 years, then odanacatib 50 mg for 8 years; participants who were treated with odanacatib 3 mg for 2 years, then odanacatib 50 mg for 8 years; and participants who were treated with odanacatib 10 mg for 2 years, then odanacatib 50 mg for 8 years.
- Group C: Odanacatib 50 mg Once Weekly: Group C consists of a combination of participants who were treated with placebo for 3 years, then odanacatib 50 mg for 7 years; and participants who were treated with odanacatib 3 mg for 2 years, then placebo for 1 year, then odanacatib 50 mg for 7 years.
- Group D: Odanacatib 50 mg Once Weekly: Group D consists of a combination of participants who were treated with odanacatib 10 mg for 2 years, then placebo for 3 years, then odanacatib 50 mg for 5 years; participants who were treated with odanacatib 25 mg for 5 years, then placebo for 3 years, then odanacatib 50 mg for 5 years; and participants who were treated with odanacatib 50 mg for 2 years, then placebo for 3 years, then odanacatib 50 mg for 5 years.
Arm/Group | Group A: Odanacatib 50 mg Once Weekly | Group B: Odanacatib 50 mg Once Weekly | Group C: Odanacatib 50 mg Once Weekly | Group D: Odanacatib 50 mg Once Weekly
Number analyzed (Participants) | 20 | 16 | 17 | 21
Percentage Change | 16.92 [12.28 to 21.55] | 14.56 [11.1 to 18.02] | 17.18 [11.48 to 22.88] | 7.71 [4.46 to 10.95]

38. Primary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE) During Treatment Years 6-10 (60 Months)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not it is considered related to the study drug.
Time Frame: Years 6-10 (up to 60 months, up to 14 days after the last dose of study drug)
Population: All participants who received at least 1 administration of the trial drug during treatment years 6-10
Measure: Number; unit: Participants
Arm/Group | Group A: Odanacatib 50 mg Once Weekly | Group B: Odanacatib 50 mg Once Weekly | Group C: Odanacatib 50 mg Once Weekly | Group D: Odanacatib 50 mg Once Weekly
Number analyzed (Participants) | 28 | 34 | 23 | 32
Participants | 27 | 34 | 23 | 32

39. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE During Treatment Years 6-10 (60 Months)
Description: as for outcome 38
Time Frame: Years 6-10 (up to 60 months)
Population: All participants who received at least 1 administration of the trial drug during treatment years 6-10.
Measure: Number; unit: Participants
Arm/Group | Group A: Odanacatib 50 mg Once Weekly | Group B: Odanacatib 50 mg Once Weekly | Group C: Odanacatib 50 mg Once Weekly | Group D: Odanacatib 50 mg Once Weekly
Number analyzed (Participants) | 28 | 34 | 23 | 32
Participants | 1 | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events data were collected up to 120 months (from start of study medication, up to 14 days after the last dose).
Description: The Safety Analysis was based on the All Participants as Treated (APaT) population, which included all participants who took at least one dose of study medication.
Groups:
- Years 1-2 Placebo/Placebo-Ext 1: One placebo tablet once a week
- Years 1-2 Odanacatib 3 mg/Odanacatib 3 Mg-Ext 1: One odanacatib 3 mg tablet once a week
- Years 1-2 Odanacatib 10 mg/Odanacatib 10 Mg-Ext 1: One odanacatib 10 mg tablet once a week
- Years 1-2 Odanacatib 25 mg/Odanacatib 25 Mg-Ext 1: One odanacatib 25 mg tablet once a week
- Years 1-2 Odanacatib 50 mg/Odanacatib 50 Mg-Ext 1: One odanacatib 50 mg tablet once a week
- Year 3 Placebo/Placebo-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one placebo tablet once a week. Before entering this extension, participants in this treatment group had taken one placebo tablet once a week for 2 years.
- Year 3 Placebo/Odanacatib 50 Mg-Ext 2: During this 12-month extension (Year 3), participants took one 50 mg tablet of odanacatib once a week. Before entering this extension, participants in this treatment group had taken one placebo tablet once a week for 2 years.
- Year 3 Odanacatib 3 mg/Placebo-Ext 2: During this 12-month extension (Year 3), participants took one placebo tablet once a week. Before entering this extension, participants in this treatment group had taken one 3 mg tablet of odanacatib once a week for 2 years.
- Year 3 Odanacatib 3 mg/Odanacatib 50 Mg-Ext 2: During this 12-month extension (Year 3), participants took one 50 mg tablet of odanacatib once a week. Before entering this extension, participants in this treatment group had taken one 3 mg tablet of odanacatib once a week for 2 years.
- Year 3 Odanacatib 10 mg/Placebo-Ext 2: During this 12-month extension (Year 3), participants took one placebo tablet once a week. Before entering this extension, participants had taken one 10 mg tablet of odanacatib once a week for 2 years.
- Year 3 Odanacatib 10 mg/Odanacatib 50 Mg-Ext 2: During this 12-month extension (Year 3), participants took one 50 mg tablet of odanacatib once a week. Before entering this extension, participants in this treatment group took one 10 mg tablet of odanacatib once a week for 2 years.
- Year 3 Odanacatib 25 mg/Placebo-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one placebo tablet once a week. Before entering this extension, participants in this treatment group had taken one 25 mg tablet of odanacatib once a week for 2 years.
- Year 3 Odanacatib 25 mg/Odanacatib 50 Mg-Ext 2: During this 12-month extension (Year 3), participants took one 50 mg tablet of odanacatib once a week. Before entering this extension, participants in this treatment group had taken one 25 mg tablet of odanacatib once a week for 2 years.
- Year 3 Odanacatib 50 mg/Placebo-Ext 2: During this 12-month extension (Year 3), participants in this treatment group took one placebo tablet once a week. Before entering this extension, participants in this treatment group had taken one 50 mg tablet of odanacatib once a week for 2 years.
- Year 3 Odanacatib 50 mg/Odanacatib 50 Mg-Ext 2: During this 12-month extension (Year 3), participants took one 50 mg tablet of odanacatib once a week. Before entering this extension, participants in this treatment group had taken one 50 mg tablet of odanacatib once a week for 2 years.
- Years 4-5 Combined Group A.1: Odanacatib 50 mg: Combined Group A.1 consists of participants who received odanacatib 50 mg once a week during Year 3.
  During this 24-month extension (Years 4-5), these participants continued to receive odanacatib 50 mg once a week.
- Years 4-5 Combined Group A.2: Odanacatib 50 mg: Combined Group A.2 consists of participants who received placebo or odanacatib 3 mg in Years 1, 2 and 3. During this 24-month extension (Years 4-5), these participants received odanacatib 50 mg once a week.
- Years 4-5 Combined Group A.3: Placebo: Combined Group A.3 consists of participants who, during this 24-month extension (Years 4-5), received placebo once a week.
- Years 6-10 Group A: Odanacatib 50 mg Once Weekly: Group A consists of a combination of participants who were treated with odanacatib 25 mg for 2 years, then odanacatib 50 mg for 8 years; and participants who were treated with odanacatib 50 mg for 10 years.
- Years 6-10 Group B: Odanacatib 50 mg Once Weekly: Group B consists of a combination participants who were treated with placebo for 2 years, then odanacatib 50 mg for 8 years; participants who were treated with odanacatib 3 mg for 2 years, then odanacatib 50 mg for 8 years; and participants who were treated with odanacatib 10 mg for 2 years, then odanacatib 50 mg for 8 years.
- Years 6-10 Group C: Odanacatib 50 mg Once Weekly: Group C consists of a combination of participants who were treated with placebo for 3 years, then odanacatib 50 mg for 7 years; and participants who were treated with odanacatib 3 mg for 2 years, then placebo for 1 year, then odanacatib 50 mg for 7 years
- Years 6-10 Group D: Odanacatib 50 mg Once Weekly: Group D consists of a combination of participants who were treated with odanacatib 10 mg for 2 years, then placebo for 3 years, then odanacatib 50 mg for 5 years; participants who were treated with odanacatib 25 mg for 5 years, then placebo for 3 years, then odanacatib 50 mg for 5 years; and participants who were treated with odanacatib 50 mg for 2 years, then placebo for 3 years, then odanacatib 50 mg for 5 years.
Arm/Group | Years 1-2 Placebo/Placebo-Ext 1 | Years 1-2 Odanacatib 3 mg/Odanacatib 3 Mg-Ext 1 | Years 1-2 Odanacatib 10 mg/Odanacatib 10 Mg-Ext 1 | Years 1-2 Odanacatib 25 mg/Odanacatib 25 Mg-Ext 1 | Years 1-2 Odanacatib 50 mg/Odanacatib 50 Mg-Ext 1 | Year 3 Placebo/Placebo-Ext 2 | Year 3 Placebo/Odanacatib 50 Mg-Ext 2 | Year 3 Odanacatib 3 mg/Placebo-Ext 2 | Year 3 Odanacatib 3 mg/Odanacatib 50 Mg-Ext 2 | Year 3 Odanacatib 10 mg/Placebo-Ext 2 | Year 3 Odanacatib 10 mg/Odanacatib 50 Mg-Ext 2 | Year 3 Odanacatib 25 mg/Placebo-Ext 2 | Year 3 Odanacatib 25 mg/Odanacatib 50 Mg-Ext 2 | Year 3 Odanacatib 50 mg/Placebo-Ext 2 | Year 3 Odanacatib 50 mg/Odanacatib 50 Mg-Ext 2 | Years 4-5 Combined Group A.1: Odanacatib 50 mg | Years 4-5 Combined Group A.2: Odanacatib 50 mg | Years 4-5 Combined Group A.3: Placebo | Years 6-10 Group A: Odanacatib 50 mg Once Weekly | Years 6-10 Group B: Odanacatib 50 mg Once Weekly | Years 6-10 Group C: Odanacatib 50 mg Once Weekly | Years 6-10 Group D: Odanacatib 50 mg Once Weekly
Serious Adverse Events (participants affected / at risk) | 8/83 | 12/82 | 10/77 | 9/79 | 14/78 | 2/19 | 2/22 | 3/18 | 2/17 | 1/18 | 1/17 | 2/19 | 3/21 | 2/18 | 1/20 | 16/73 | 2/27 | 8/41 | 8/28 | 14/34 | 6/23 | 12/32
Other Adverse Events (participants affected / at risk) | 68/83 | 66/82 | 67/77 | 67/79 | 66/78 | 17/19 | 13/22 | 16/18 | 14/17 | 13/18 | 15/17 | 15/19 | 17/21 | 14/18 | 15/20 | 64/73 | 24/27 | 33/41 | 25/28 | 31/34 | 23/23 | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Years 1-2 Placebo/Placebo-Ext 1 (N=83) | Years 1-2 Odanacatib 3 mg/Odanacatib 3 Mg-Ext 1 (N=82) | Years 1-2 Odanacatib 10 mg/Odanacatib 10 Mg-Ext 1 (N=77) | Years 1-2 Odanacatib 25 mg/Odanacatib 25 Mg-Ext 1 (N=79) | Years 1-2 Odanacatib 50 mg/Odanacatib 50 Mg-Ext 1 (N=78) | Year 3 Placebo/Placebo-Ext 2 (N=19) | Year 3 Placebo/Odanacatib 50 Mg-Ext 2 (N=22) | Year 3 Odanacatib 3 mg/Placebo-Ext 2 (N=18) | Year 3 Odanacatib 3 mg/Odanacatib 50 Mg-Ext 2 (N=17) | Year 3 Odanacatib 10 mg/Placebo-Ext 2 (N=18) | Year 3 Odanacatib 10 mg/Odanacatib 50 Mg-Ext 2 (N=17) | Year 3 Odanacatib 25 mg/Placebo-Ext 2 (N=19) | Year 3 Odanacatib 25 mg/Odanacatib 50 Mg-Ext 2 (N=21) | Year 3 Odanacatib 50 mg/Placebo-Ext 2 (N=18) | Year 3 Odanacatib 50 mg/Odanacatib 50 Mg-Ext 2 (N=20) | Years 4-5 Combined Group A.1: Odanacatib 50 mg (N=73) | Years 4-5 Combined Group A.2: Odanacatib 50 mg (N=27) | Years 4-5 Combined Group A.3: Placebo (N=41) | Years 6-10 Group A: Odanacatib 50 mg Once Weekly (N=28) | Years 6-10 Group B: Odanacatib 50 mg Once Weekly (N=34) | Years 6-10 Group C: Odanacatib 50 mg Once Weekly (N=23) | Years 6-10 Group D: Odanacatib 50 mg Once Weekly (N=32)
Arteriospasm Coronary (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary Artery Occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoparathyroidism secondary (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular Hole (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal Detachment (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal Fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post Procedural Bile Leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram ST-T Change (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (5) | 1 (1) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast Cancer In Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Reversible Ischaemic Neurological Deficit (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital Prolapse (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIIth Nerve Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal Sphincter Atony (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurilemmoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nerve root compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Years 1-2 Placebo/Placebo-Ext 1 (N=83) | Years 1-2 Odanacatib 3 mg/Odanacatib 3 Mg-Ext 1 (N=82) | Years 1-2 Odanacatib 10 mg/Odanacatib 10 Mg-Ext 1 (N=77) | Years 1-2 Odanacatib 25 mg/Odanacatib 25 Mg-Ext 1 (N=79) | Years 1-2 Odanacatib 50 mg/Odanacatib 50 Mg-Ext 1 (N=78) | Year 3 Placebo/Placebo-Ext 2 (N=19) | Year 3 Placebo/Odanacatib 50 Mg-Ext 2 (N=22) | Year 3 Odanacatib 3 mg/Placebo-Ext 2 (N=18) | Year 3 Odanacatib 3 mg/Odanacatib 50 Mg-Ext 2 (N=17) | Year 3 Odanacatib 10 mg/Placebo-Ext 2 (N=18) | Year 3 Odanacatib 10 mg/Odanacatib 50 Mg-Ext 2 (N=17) | Year 3 Odanacatib 25 mg/Placebo-Ext 2 (N=19) | Year 3 Odanacatib 25 mg/Odanacatib 50 Mg-Ext 2 (N=21) | Year 3 Odanacatib 50 mg/Placebo-Ext 2 (N=18) | Year 3 Odanacatib 50 mg/Odanacatib 50 Mg-Ext 2 (N=20) | Years 4-5 Combined Group A.1: Odanacatib 50 mg (N=73) | Years 4-5 Combined Group A.2: Odanacatib 50 mg (N=27) | Years 4-5 Combined Group A.3: Placebo (N=41) | Years 6-10 Group A: Odanacatib 50 mg Once Weekly (N=28) | Years 6-10 Group B: Odanacatib 50 mg Once Weekly (N=34) | Years 6-10 Group C: Odanacatib 50 mg Once Weekly (N=23) | Years 6-10 Group D: Odanacatib 50 mg Once Weekly (N=32)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (4) | 3 (3) | 0 (0) | 6 (9) | 6 (10) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 5 (5) | 5 (5) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 8 (8) | 6 (7) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 1 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 4 (5) | 8 (8) | 3 (3) | 7 (10) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (3) | 3 (3) | 0 (0) | 2 (2) | 2 (3) | 4 (5) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 4 (6) | 2 (3) | 3 (4) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 3 (3)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4) | 5 (7) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (8) | 4 (6) | 6 (7) | 6 (7) | 5 (7) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (7) | 3 (4) | 4 (6) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 6 (6) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza Like Illness (General disorders) | 3 (3) | 1 (1) | 3 (5) | 2 (2) | 6 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (5) | 4 (6) | 4 (5) | 2 (2) | 1 (2) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (7) | 4 (4) | 4 (4) | 3 (4) | 5 (6) | 5 (9) | 5 (5)
Cystitis (Infections and infestations) | 1 (3) | 6 (6) | 3 (3) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (4) | 2 (3) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4) | 4 (4) | 5 (6) | 4 (5) | 5 (6) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (5) | 2 (2) | 1 (1) | 1 (2) | 4 (4) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 9 (11) | 10 (12) | 7 (9) | 7 (11) | 10 (14) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 2 (7) | 3 (5) | 2 (2) | 2
Urinary Tract Infection (Infections and infestations) | 11 (17) | 6 (7) | 7 (7) | 8 (10) | 12 (15) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 10 (12) | 4 (4) | 2 (3) | 9 (15) | 9 (19) | 6 (20) | 7 (15)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 2 (4) | 5 (8) | 2 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (2) | 3 (7)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 3 (4) | 0 (0) | 5 (7) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 3 (5) | 2 (2) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Weight Decreased (Investigations) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 2 (2)
Weight Increased (Investigations) | 4 (4) | 2 (2) | 3 (3) | 5 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (24) | 12 (16) | 12 (13) | 14 (17) | 12 (14) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 3 (4) | 0 (0) | 3 (4) | 9 (13) | 4 (4) | 6 (8) | 5 (10) | 4 (4) | 8 (8) | 3 (3)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7) | 7 (7) | 3 (3) | 13 (16) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 5 (5) | 10 (11) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 4 (5) | 1 (1) | 6 (6) | 3 (6) | 4 (4) | 5 (6) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 4 (4) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 3 (4) | 3 (4) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 4 (5) | 4 (4) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 6 (7) | 2 (3) | 1 (2) | 3 (3) | 5 (6) | 2 (2) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 4 (5) | 7 (9) | 8 (10) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 11 (13) | 9 (9) | 10 (10) | 9 (10) | 9 (12) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 1 (1) | 2 (3) | 3 (4) | 3 (4)
Depression (Psychiatric disorders) | 5 (5) | 4 (4) | 5 (5) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 4 (5) | 2 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 7 (7) | 3 (4) | 4 (4) | 3 (3) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 7 (10) | 4 (4) | 5 (6) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 7 (7) | 3 (3) | 8 (8) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 5 (6) | 2 (2) | 2 (2) | 3 (3) | 6 (7) | 5 (5) | 3 (3)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral Valve Prolapse (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Tympanosclerosis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 4 (5) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
Thyroiditis Chronic (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis Allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular Degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Anal Fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Duodenal Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecal Incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric Polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Gingival Swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Calcinosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 4 (8) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 2 (3) | 0 (0)
Allergy To Arthropod Sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Eye Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fungal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 5 (7)
Nasal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 14 (20) | 9 (13) | 16 (20) | 8 (10) | 14 (23) | 1 (1) | 4 (5) | 2 (3) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (2) | 13 (16) | 6 (13) | 10 (13) | 7 (9) | 8 (15) | 5 (9) | 9 (20)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 1 (2)
Oral Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2)
Otitis Media Acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (3) | 1 (1) | 3 (4)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthropod Sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 3 (13) | 4 (8) | 5 (6) | 4 (9)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 2 (2) | 3 (3) | 3 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull Fractured Base (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood 1,25-Dihydroxycholecalciferol Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Cholesterol Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Glucose Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1
Blood Parathyroid Hormone Increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (13) | 3 (5) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Triglycerides Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid Bruit (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose Urine Present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
High Density Lipoprotein Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White Blood Cells Urine Positive (Investigations) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 4 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 10 (12) | 17 (19) | 9 (11) | 14 (19) | 11 (13) | 2 (2) | 5 (5) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 8 (11) | 5 (7) | 1 (1) | 6 (6) | 7 (9) | 5 (7) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 10 (13) | 8 (10) | 8 (8) | 11 (11) | 3 (5) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 12 (15) | 4 (5) | 2 (2) | 6 (6) | 1 (1) | 2 (3) | 7 (9)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 2 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigeminal Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dysthymic Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Breast Mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fibrocystic Breast Disease (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal Discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (2) | 2 (5) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (4)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Granuloma Annulare (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichen Planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sebaceous Hyperplasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicose Vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eyelid Ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.